CLINICAL TRIAL: NCT06765148
Title: Radiodiagnostic Properties of Maxillary Antroliths: a Retrospective Cone Beam Computed Tomography Study
Brief Title: Radiodiagnostic Properties of Maxillary Antroliths
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, DİLARA NİL GÜNAÇAR, Assoc. Prof., Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 2024/299
Record Dates: First submitted 2024-12-24; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Antrolith; Maxillary Sinus
Keywords: cone beam computed tomography; Lithiasis; maxillary sinus; panoramic radiography
MeSH Terms: conditions — Lithiasis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Retrospective radiologic study — Retrospective radiologic study

SUMMARY:
Background: To evaluate the frequency and radiodiagnostic characteristics of maxillary antroliths using cone beam computed tomography.

Materials and Methods: A review of 1166 patients aged 11-85 years was conducted to assess the frequency of maxillary antroliths, considering sex, age, and location. The relationship between antroliths and sex, location, dental treatment status, and sinus inflammation was evaluated. The shape, size, and volume of the antroliths were also analyzed. Significance was set at p=0.05 for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* DPR and CBCT and also had a maximum of 3 months
* Image quality was sufficient
* No artifacts CBCT images

Exclusion Criteria:

* Tomographic images that contained pathologies such as cysts/tumors in the
* Insufficient diagnostic quality
* History of maxillofacial trauma or surgery, any syndrome/bone-related disease/metabolic disease
* Insufficient diagnostic quality or patient position-related artifacts

Ages: 11 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective maxillary sinus included CBCT images
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2024-12-22 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Antrolith descriptive analysis | for three days from the beginning of the study
  CBCT images were examined in axial, sagittal, and coronal slices to investigate the presence of antroliths. The age and sex information of the detected cases were recorded.
Antrolith localization and relationship the dental status evaluation | for three days from the beginning of the study
  Each sinus cavity exhibiting antroliths was evaluated for distribution and location as follows: (1) unilateral or bilateral, (2) single or multiple, (3) tooth extraction/root canal treatment/residual root fragment/implant/periodontal disease and/or periapical lesion (any dental cause of sinus inflammation), (4) premolar or molar region, and (5) sinus floor, lateral wall, or medial wall.
Antrolith and mucosal thickness classification | for three days from the beginning of the study
  the detected antroliths were categorized according to the classification of Cho et al. In this classification made according to the sizes of antroliths, Punctate = ≤3 mm in both height and width, Linear = ≤3 mm and more than treble in width, and Amorphous = >3 mm in both width and height.
  Additionally, the locations of the openings of the maxillary sinus ostiums were evaluated, and mucosal thickening, if any, was measured. Mucosal thickness measurements were made on coronal slices using NewTom's NNT viewer measuring tool. Similar to Chen et al., the sinus membrane thickness was measured perpendicular to the bone wall, from the maximum thickest region. Similar to Chen et al.'s classification of sinus membrane thickness measurements, which used Block and Dostoury's classification, the mucosal thickness was classified into three subgroups: membrane thicknesses <2 mm, 2-5 mm, and >5 mm. Also, similar to the article by Cho et al., the degree of inflammation in the maxillary sinus was
Antrolith volume measurement | for three days from the beginning of the study
  3D reconstruction and volume measurements of antroliths were performed using the ITK SNAP software (free software under the GNU General Public License developed by the National Institutes of Health, the US National Institute of Biomedical Imaging and Bioenergy needs, the US National Library of Medicine, the Universities of Pennsylvania and North Carolina, and an independent group of developers).
Different images evaluation for antrolit | for three days from the beginning of the study
  In addition, the visibility of antroliths detected on CBCT was also evaluated using panoramic radiographs taken from the patient (Fig 2). The detectability of antroliths in DPRs was evaluated by observers as detectable, suspicious, and undetectable.

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdogan University Training and Research Hospital, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gunacar DN, Kose TE, Ceren F. Radiodiagnostic properties of maxillary antroliths: a retrospective cone beam computed tomography study. BMC Oral Health. 2025 Feb 19;25(1):259. doi: 10.1186/s12903-025-05641-y. PMID 39972501